CLINICAL TRIAL: NCT02738463
Title: Role of Maternal Serum Ferritin in the Prediction of Low Neonatal Birth Weight
Brief Title: Maternal Serum Ferritin and Low Neonatal Birth Weight
Acronym: LBW
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa Mahmoud salem, principal investigator, Ain Shams Maternity Hospital
Other Study IDs: SHMS1985
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: IUGR
Keywords: ferritin LBW

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 case: This group will include 32 pregnant females whose fetuses show intrauterine growth restriction at full term ( the 32 neonates with birth weight less than 10th percentile for corresponding gestational age will be included as small for gestational age and the investigator will thaw their maternal frozen samples for detection of serum ferritin level)
- Group 2 control: This group will include at least 32 pregnant females whose fetuses are appropriate for gestational age at full term ( the 32 neonates with birth more than or equal to the 10th percentile for corresponding gestational age will be included as average for gestational age and the investigator will thaw their maternal frozen samples for detection of serum ferritin level)

SUMMARY:
Intrauterine growth restriction ( IUGR )is defined as fetal growth slower than the normal growth potential of a specific fetus because of genetic or environmental factors. Recently several studies have highlighted the role of many biomolecules as markers for IUGR. Measurement of maternal serum ferritin has also been used as a predictive marker for increased risk of IUGR. Iron deficiency has its known deleterious effect in pregnancy but iron loading may be associated with oxidative damage to cells and tissues. It has been shown in various studies that lower level of transferritin receptor expression in placenta is associated with preeclampsia and IUGR. This can lead to decrease extraction of iron by placenta from maternal serum leading to increase maternal serum ferritin. This fetal iron deficiency leads to increase in fetal corticotropins and fetal cortisol, causing inhibition of fetal growth

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) is defined as fetal growth slower than the normal growth potential of a specific fetus because of genetic or environmental factors. IUGR is associated with a high incidence of perinatal morbidity and mortality. IUGR neonates have a greater risk of hypoxic ischemic encephalopathy, intraventricular hemorrhage and necrotizing enterocolitis with longer hospital stay and higher health care costs. Incidence of a fetus developing a small size for gestational age is about 8%. Fetal growth is regulated by the balance between fetal nutrient demand and maternal placental nutrient supply. Intrauterine growth restriction may be caused by maternal, placental, or fetal factors. Nearly one-third of IUGRs are due to genetic causes, and two-thirds are related to the fetal environment. In the developing world, IUGR is likely to be a consequence of poor maternal nutritional status prior to or during pregnancy.

There are two general patterns of growth abnormalities: symmetric and asymmetric. Symmetric growth inhibition arises during the first half of gestation, when fetal growth occurs primarily through cellular division and produces an undersized fetus with fewer cells of normal size. Asymmetric growth inhibition occurs during the second half of gestation and is usually the consequence of an inadequate availability of substrates for fetal metabolism. To prevent the previously mentioned complications of IUGR, it is important to establish markers which can identify pregnancies at risk of IUGR early enough. Recently several studies have highlighted the role of many bio-molecules as markers for IUGR like leptin, adiponectin, endothelin-1, lactate dehydrogenase, s-endoglin, pregnancy associated plasma protein, metastin. Apart from being expensive, laboratories at majority of centers are not equipped with facilities of measurement of these markers. Measurement of maternal serum ferritin has also been used as a predictive marker for increased risk of IUGR in one previous study on a limited number (seventeen) of cases. Ferritin is an intracellular protein consisting of 24 heavy and light sub-units surrounding a core that can store up to 4,500 iron atoms. The two sub-units are highly conserved during evolution, but only the heavy sub-unit has ferroxidase activity. Ferritin is released by infiltrating leukocytes, in response to acute and chronic infection. Ferritin as an acute phase reactant is well known for its intracellular iron sequestration and storage abilities during immune activation. Serum ferritin concentration is positively correlated with the amount of total body iron stores in the absence of inflammation. Serum ferritin is considered a valuable bio-marker for body iron status in healthy subjects.Iron deficiency has its known deleterious effect in pregnancy but iron loading may be associated with oxidative damage to cells and tissues. It has been shown in various studies that lower level of transferritin receptor expression in placenta is associated with preeclampsia and IUGR. This can lead to decrease extraction of iron by placenta from maternal serum leading to increase maternal serum ferritin. This fetal iron deficiency leads to increase in fetal corticotropins and fetal cortisol, causing inhibition of fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years of age
* Pregnant with singleton intrauterine pregnancy
* 30th-32nd weeks of gestation

Exclusion Criteria:

* Patients with a history of anemia due to any causes.
* Patients with history of iron supplementation, Clinical and/or laboratory evidence of hepatic, renal, hematologic, cardiovascular abnormalities.
* History of acid-peptic disorders, esophagitis, or hiatal hernia.
* Family history of thalassemia, sickle cell anemia, or malabsorption syndrome.
* Antepartum hemorrhage.
* Allergies to milk proteins / hypersensitivity to iron preparations.
* Patients with acute infection, positive CRP, raised TLC count.
* Congenital malformation and fetuses with chromosomal or genetic syndrome.
* Recent blood transfusion.
* Refusal to participate in the study.
* BMI <18.
* Placental abnormalities like velamentous insertion.
* Multiple pregnancies.
* Smoking during pregnancy
* Preterm births.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include women, who attend the Obstetrics Department, in Ain Shams University Hospital, and fulfill the inclusion criteria, after taking an informed consent
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
maternal serum ferritin (microg/L) | 2 months
  Ferritin values will be estimated by immunometric testing for quantitative determination in human serum at Olympus analyzers using the Olympus ferritin reagent. Reference ranges from 10.00 to 30.00 microgram/L
Fetal weight (gm) | 5 minutes
  birth weight less than 10th percentile will be adjusted for small for gestational age

SECONDARY OUTCOMES:
Maternal hemoglobin (g/L) | 2 months
  estimation will be done from hemolysate of the obtained blood samples with the addition of sodium ferricyanide and sodium cyanide. Cyanmet -hemoglobin formed in the solution will be estimated by spectro photometry at the wave length of 540 nm.
Maternal hematocrit (x10^12/L) | 2 months
  The level will be also estimated by spectro photometry and calculated using the following formula: Hematocrit = blood cells volume/volume of blood sample × 100.
Apgar score | 5 minutes
  will be estimated by cardiac action, respiration of the newborn, muscle tone, skin color and reaction of the newborn will be estimated by 0, 1 or 2 summed up and compared. Apgar score can vary from 0 to 10.
Maternal total leucocytic count (x10^9/L) | 2 months
  will be also estimated also by spectro photometry

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Bayoumyi, MD, Study Chair — Ain Shams University; Sherif A Ashoush, MD, Study Director — Ain Shams University; Haitham AM ElSabaa, MD, Study Director — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams Maternity Hospital, Cairo, Cairo Governorate
  - outpatient clinics in the Obstetrics and Gynecology Department Ain Shams Maternity Hospital, Cairo, Cairo Governorate

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Arosio P, Ingrassia R, Cavadini P. Ferritins: a family of molecules for iron storage, antioxidation and more. Biochim Biophys Acta. 2009 Jul;1790(7):589-99. doi: 10.1016/j.bbagen.2008.09.004. Epub 2008 Sep 26. PMID 18929623
- [Background] Bindal N, Godha Z, Kohli R, Kadam VK. Role of maternal serum ferritin as a predictive marker in intrauterine growth restriction. Int J Reprod Contracept Obstet Gynecol. 2015 Jun;4(3):804-808
- [Background] Milman N. Iron Deficiency and Anaemia in Pregnant Women in Malaysia - Still a Significant and Challenging Health Problem. J Preg Child Health 2015, 2:3
- [Background] Moh W, Graham JM Jr, Wadhawan I, Sanchez-Lara PA. Extrinsic factors influencing fetal deformations and intrauterine growth restriction. J Pregnancy. 2012;2012:750485. doi: 10.1155/2012/750485. Epub 2012 Jul 19. PMID 22888434
- [Background] Murki S and Sharma D. Intrauterine Growth Retardation - A Review Article. Murki and Sharma, J Neonatal Biol 2014, 3:3
- [Background] Nandini M D, Shetty HV, Rupakala BV, Usha S M R, Priyadarshini KS, Manjula HS and Victoria Ksh. Study of serum ferritin levels in preterm labor. International Journal of Recent Trends in Science and Technology, ISSN 2277-2812 E-ISSN 2249-8109, Volume 14, Issue 2, 2015 pp 477-480
- [Background] Muhammad T, Khattak AA, Shafiq-ur-Rehman, Khan MA, Khan A, Khan MA. Maternal factors associated with intrauterine growth restriction. J Ayub Med Coll Abbottabad. 2010 Oct-Dec;22(4):64-9. PMID 22455264
- [Background] Višnjevac N, Segedi LM, Ćurčić A, Višnjevac J, Dragan Stajić. Blood ferritin levels in pregnant women and prediction of the development of fetal intrauterine growth restriction. J Med Biochem. 2011;30:m317-22
- [Background] Wang CN, Chang SD, Peng HH, Lee YS, Chang YL, Cheng PJ, Chao AS, Wang TH, Wang HS. Change in amniotic fluid levels of multiple anti-angiogenic proteins before development of preeclampsia and intrauterine growth restriction. J Clin Endocrinol Metab. 2010 Mar;95(3):1431-41. doi: 10.1210/jc.2009-1954. Epub 2010 Jan 15. PMID 20080845
- [Background] Zhang S, Regnault TR, Barker PL, Botting KJ, McMillen IC, McMillan CM, Roberts CT, Morrison JL. Placental adaptations in growth restriction. Nutrients. 2015 Jan 8;7(1):360-89. doi: 10.3390/nu7010360. PMID 25580812
- See also: Ross MG. Fetal growth restriction, 2008 — http://emedicine.medscape.com/article/261226-overview
- Available data/document: Individual Participant Data Set — http://www.ncbi.nlm.nih.gov/pubmed